CLINICAL TRIAL: NCT05882604
Title: Treatment of Temporomandibular Joint Internal Derangement Using MESNA Injection
Brief Title: MESNA Injection for TMJ Internal Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdellatif Abdelfatah, Lecturer of oral and maxillofacial surgery, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #R-OS-4-23-3
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Mesna; Arthrocentesis; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-articular injection with MESNA solution (Experimental): 1 ml of MESNA will be injected intra-articular
  Interventions: Drug: Mesna Injection
- Arthrocentesis with ringer solution (Active Comparator): ringer solution will be used for arthrocentesis
  Interventions: Drug: Arthrocentesis with ringer solution

INTERVENTIONS:
Drug: Mesna Injection — 1 ml of MESNA will be injected using 20-guage needle in he upper compartment of TMJ in patient with internal derrangement.
  Arms: Intra-articular injection with MESNA solution
Drug: Arthrocentesis with ringer solution — Two 20-gauge needles will be placed into upper joint space as entry and exit points for washing.The arthrocentesis will be performed with 100 ml of lactated Ringer's solution to eliminate the inflammatory mediators present in the synovial fluid
  Arms: Arthrocentesis with ringer solution

SUMMARY:
The pathogenesis of temporomandibular disorders focusing on the biochemistry of the synovial fluid in various stages of temporomandibular joint disease. The role of inflammation has been investigated and proposed as an underlying mechanism of pain and dysfunction of temporomandibular joint. MESNA (sodium 2-mercaptoethanesulfonate) was approved several years ago and marketed in several formulations as a mucolytic agent in the respiratory field, since it breaks the disulfide bonds between polypeptide chains of mucus. The tissue distribution of MESNA is negligible, and the elimination of the substance is rapidly and completely achieved by kidney

DETAILED DESCRIPTION:
Clarification (July 2025): Recruitment was completed in March 2023 following clinical scheduling and preliminary departmental clearance, while formal written ethical approval was finalized in early April 2023. All patients were followed up for one year, and the study was completed by March 2024.

ELIGIBILITY:
Inclusion Criteria:

* patients with TMJ internal derangement with reduction

Exclusion Criteria:

* inflammatory or connective tissue disease
* autoimmune disease history
* neurologic problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
maximal interincisal opening (MIO) | 6 months
  a digital caliper will be employed to measure the maximum interincisal opening pre and postoperative

SECONDARY OUTCOMES:
Joint pain | 6 months
  pain will be assessed on a visual analogue scale (VAS) with a score between 0 and 10, 0 means no pain and 10 means severe pain
clicking sound | 6 months
  yes or no questionnaire,yes mean clicking is present and no means clicking disappeared

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No